CLINICAL TRIAL: NCT02738125
Title: Assessing Effectiveness of Adalimumab for Treating Ulcerative Colitis in Real Life Conditions
Acronym: SOTHIS
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-681
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Adalimumab; Ulcerative Colitis; SOTHIS; Effectiveness
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects starting/ receiving adalimumab: Subjects starting/ receiving Adalimumab for UC

SUMMARY:
This study assesses the long?term effectiveness of adalimumab in subjects starting a treatment for ulcerative colitis in real life conditions, namely to describe the time to loss of clinical benefit in a time to event approach.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from ulcerative colitis
* Naïve from Adalimumab
* Starting a treatment with adalimumab
* Capable of and willing to grant authorization for use/disclosure of data collected
* Able to read, understand, and complete patients questionnaires

Exclusion Criteria:

- None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects starting/ receiving Adalimumab for UC
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Time to loss of clinical benefit | Up to Month 120
  Loss of clinical benefit will be defined as one of the following: loss of efficacy leading to adalimumab discontinuation or introduction/reinforcement of aminosalicylates, 6-mercaptopurine, or azathioprine, introduction or reinforcement of corticosteroids (any route), UC-related surgery, discontinuation of adalimumab due to adverse event, death.

SECONDARY OUTCOMES:
Change from Baseline (Month 0) in Steroid-free remission | From Month 0 to Month 120
  Steroid- free remission is defined as partial Mayo score <= 2 with no subscore >1 and no daily intake of prednisone.
Change from Baseline (Month 0) in Clinical Remission | From Month 0 to Month 120
  Clinical remission is defined as partial Mayo score <= 2 with no subscore >1
Change from Baseline (Month 0) in Clinical Response | From Month 0 to Month 120
  Clinical response is decrease in partial Mayo score >= 3 points and >= 30% from baseline plus a decrease in rectal bleeding subscore >= 1 or an absolute rectal bleeding subscore <= 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (80):
- France (80):
  - Chu de Nice-Hopital L'Archet Ii /Id# 151132, Nice, Alpes-Maritimes
  - Chu de Nice-Hopital L'Archet Ii /Id# 151181, Nice, Alpes-Maritimes
  - CHU Clermont-Ferrand /ID# 153527, Clermont, Auvergne-Rhône-Alpes
  - HCL - Hôpital Lyon Sud /ID# 151146, Pierre-Bénite, Auvergne-Rhône-Alpes
  - HCL - Hôpital Lyon Sud /ID# 151505, Pierre-Bénite, Auvergne-Rhône-Alpes
  - HCL - Hôpital Lyon Sud /ID# 165859, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hopital Saint Joseph /ID# 164405, Marseille, Bouches-du-Rhone
  - APHM - Hopital Nord /ID# 152620, Marseille, Bouches-du-Rhone
  - CHU NIMES - Hopital Caremeau /ID# 169178, Nîmes, Gard
  - Cabinet Medical /ID# 155460, BAIE Mahault, Guadeloupe
  - CHU Toulouse - Hopital Purpan /ID# 167179, Toulouse, Haute-Garonne
  - CH Annecy Genevois Site Annecy /ID# 151131, Pringy, Haute-Savoie
  - CHRU Lille - Hopital Claude Huriez /ID# 151514, Lille, Hauts-de-France
  - CHRU Nancy - Hôpitaux de Brabois /ID# 151147, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 166807, Saint Priest EN Jarez, Pays de la Loire Region
  - CH Henri Duffaut /ID# 151383, Avignon, Provence-Alpes-Côte d'Azur Region
  - CH Henri Duffaut /ID# 151499, Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Cote /ID# 163714, Bayonne, Pyrenees-Atlantiques
  - Centre Hosp Intercommunal de Creteil /ID# 152361, Créteil, Val-de-Marne
  - Centre Medical Alexandre Dumas /Id# 165857, Amiens
  - Duplicate_Hopital Robert Ballanger /ID# 151382, Aulnay-sous-Bois
  - Polyclinique du Tondu /ID# 161977, Bordeaux
  - Centre Endo Nord Isere /ID# 151390, Bourgoin
  - Geier, Cabinet Medical /ID# 149652, Brest
  - Hopital de la Cavale Blanche /ID# 152618, Brest
  - Hopital de la Cavale Blanche /ID# 153608, Brest
  - Cabinet Medical /ID# 151391, Caen
  - CHRU Tours - Hopital Trousseau /ID# 163503, Chambray-lès-Tours
  - Pole Sante Leonard de Vinci /ID# 151384, Chambray-lès-Tours
  - Ch Chauny /Id# 151149, Chauny
  - CH du Haut Anjou /ID# 151151, Château-Gontier
  - Hopital Louis Mourier,Colombes /ID# 152650, Colombe
  - GHPSO CH Creil /ID# 151117, Creil
  - Cabinet Medical /ID# 150978, Douarnenez
  - Cabinet Medical /ID# 150845, Erstein
  - Centre Gastro Loire /ID# 151387, Gien
  - Clinique du Palais /ID# 151175, Grasse
  - CH La Rochelle - Hopital Saint Louis /ID# 151182, La Rochelle
  - CHU Grenoble - Hopital Michallon /ID# 151508, La Tronche
  - Duplicate_HOPITAL DUPUYTREN /ID# 157889, Limoges
  - CH Des Deux Vallees Longumeau /ID# 150977, Longjumeau
  - HCL - Hopital Edouard Herriot /ID# 151513, Lyon
  - Centre des consultations spécialisées de la sauvegarde /ID# 151515, Lyon
  - Centre Medical Les Sources /ID# 151174, Montigny-lès-Cormeilles
  - AP-HP - Hopital Saint-Louis /ID# 151509, Paris
  - Hopital Paris Saint-Joseph /ID# 153526, Paris
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 151176, Paris
  - Cabinet Medical /ID# 151118, Paris
  - Cabinet Medical /ID# 152362, Paris
  - Duplicate_CHU LYON SUD /ID# 153801, Pierre-Bénite
  - Cabinet Medical /ID# 151092, Plérin
  - Cabinet Medical /ID# 151093, Plérin
  - Cabinet Medical /ID# 151094, Plérin
  - Cabinet Medical /ID# 151148, Poissy
  - Cabinet Medical /ID# 151555, Prades-le-Lez
  - CHRU Pontchaillou /ID# 166806, Rennes
  - CHU La Réunion - site St Denis - Félix-Guyon /ID# 151556, Saint-Denis
  - Centre de Consultations /ID# 151128, Saint-Nazaire
  - Centre de Consultations /ID# 151164, Saint-Nazaire
  - Centre de Consultations /ID# 155458, Saint-Nazaire
  - Cabinet Medical /ID# 151559, Saint-Quentin
  - CHU d'Amiens /ID# 152651, Salouël
  - Cabinet Medical /ID# 151558, Saverne
  - Cabinet Medical /ID# 151162, Strasbourg
  - Centre Medical du Clos de Pacy /ID# 151129, Sucy-en-Brie
  - Maison de Santé Protestante Bordeaux Bagatelle /ID# 151497, Talence
  - Cabinet Medical, Dr. Constant, /ID# 151119, Toulon
  - Clinique Pasteur /ID# 151088, Toulouse
  - Clinique Pasteur /ID# 155792, Toulouse
  - Clinique Ambroise Pare /ID# 161978, Toulouse
  - Cabinet Medical /ID# 170136, Toulouse
  - Cabinet Medical /ID# 152841, Toulouse
  - CHU Toulouse - Hopital Rangueil /ID# 157890, Toulouse
  - Duplicate_Hopital Trousseau /ID# 150168, Tours
  - Cabinet Medical /ID# 151557, Troyes
  - GH Mutualiste Les Portes Du Sud /ID# 152374, Vénissieux
  - GH Mutualiste Les Portes Du Sud /ID# 159231, Vénissieux
  - Centre Hépato-Biliaire - Hopital Paul-Brousse /ID# 151152, Villejuif
  - Cabinet Medical /ID# 152617, Voiron
  - Hopital Beaujon /ID# 151498, Clichy, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P15-681#additional-resources-section